CLINICAL TRIAL: NCT03326609
Title: Local Anesthetic Concentration and Nerve Block Duration: A Randomized, Blinded Study in Healthy Volunteers
Brief Title: Local Anesthetic Concentration and Nerve Block Duration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Innovation Fund Denmark (Individual)
Responsible Party: Principal Investigator, Claus Behrend Christiansen, Medical doctor, Nordsjaellands Hospital
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-17022555
Record Dates: First submitted 2017-09-29; First posted 2017-10-31 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Peripheral Nerve Block
MeSH Terms: interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Volume: 2.5 mL (Experimental): Perineural injection of ropivacaine 10 mg, 2.5 mL. Concentration: Ropivacaine 4 mg/mL.
  Interventions: Drug: Ropivacaine
- Volume: 5 mL (Experimental): Perineural injection of ropivacaine 10 mg, 5 mL. Concentration: Ropivacaine 2 mg/mL
  Interventions: Drug: Ropivacaine
- Volume: 10 mL (Experimental): Perineural injection of ropivacaine 10 mg, 10 mL Concentration: Ropivacaine 1 mg/mL
  Interventions: Drug: Ropivacaine
- Volume: 15 mL (Experimental): Perineural injection of ropivacaine 10 mg, 15mL Concentration: Ropivacaine 0.67 mg/mL
  Interventions: Drug: Ropivacaine
- Volume: 20 mL (Experimental): Perineural injection of ropivacaine 10 mg, 20mL Concentration: Ropivacaine 0.5 mg/mL
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Perineural injection using a peripheral nerve block catheter and a constant infusion rate (10mL/h)
  Other Names: Isotonic saline (natriumchloride)

SUMMARY:
Background: Local anesthetic (LA) concentration and nerve block duration is sparsely described in a heterogenic study mass.

Aim: To investigate the effect of LA concentration on peripheral nerve block duration in healthy volunteers.

Methods: Randomization of 60 healthy volunteers who will receive 1 of 5 different volumes of LA (ropivacaine) using a constant dose.

Primary endpoint: Sensory nerve block defined by insensitivity towards cold.

DETAILED DESCRIPTION:
Background:

Important factors for a safe and successful nerve block include volume, dose and concentration of local anesthetic (LA). Knowing the duration of peripheral nerve blocks is important to prevent pain breakthrough. With the advancements in ultrasound (US)-guided nerve block techniques it has been possible to substantially reduce the amount of LA required to perform a successful nerve block. This has reduced the risk of systemic toxicity. However, lowering LA volume may reduce nerve block duration, but the extent of this is sparsely described in a heterogenic study mass.

Diluted and large volumes of LA seem to correlate with nerve block duration. Furthermore, increasing LA concentration seems to increase the level of motor block, but not the block duration. A long-lasting nerve block without dense motor block is preferable for optimized pain control and better opportunities to rehabilitate/ambulate.

Aim:

To investigate the effect of LA concentration on common peroneal nerve block duration in healthy volunteers.

Methods:

Randomization of 60 healthy volunteers who will receive 1 of 5 different volumes of LA (ropivacaine) using a constant dose (10mg).

Primary outcome: Duration of sensory nerve block defined by insensitivity towards cold.

Secondary outcome: Duration of motor nerve block defined by either paresis or paralysis.

Explorative outcomes: Degrees of sensory and motor nerve block; Onset times of sensory and motor nerve block; Length of neural exposure to LA.

ELIGIBILITY:
Inclusion criteria

1. Male or female from and above 18 years of age
2. ASA classification ≤ II

Exclusion criteria

1. BMI below 18 kg/m2
2. Former surgery to the lower extremity in which intervention is planned and surgery which may have caused neural damage to the common peroneal nerve/affected the sensory distribution area of the common peroneal nerve
3. Peripheral nerve disease
4. Allergy to LA
5. Pregnancy or breastfeeding
6. Enrolment in other investigational drug studies or recent clinical trials that may interfere with this study
7. Habitual use of any kind of analgesic treatment
8. Anatomic abnormalities preventing successful US-guided peripheral nerve catheter insertion

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2018-01-05 (Actual)

PRIMARY OUTCOMES:
Duration of sensory nerve block | 1-24 hours
  Insensitivity towards cold. Testing will start after onset of sensory nerve block and will be done in intervals of 60 minutes hereafter and continue until return of normal sensation.

SECONDARY OUTCOMES:
Duration of motor nerve block | 1-24 hours
  Paresis or paralysis of ankle dorsiflexion. Testing will start after onset of sensory nerve block and will be done in intervals of 60 minutes hereafter and continue until return of normal sensation.

OTHER OUTCOMES:
Length of neural exposure to local anesthetic | 10 minutes
  Ultrasound-guided measurement of the perineural spread of local anesthetic. From the most distal to the most proximal point. Measured in millimetres.
Onset of sensory nerve block | 10-180 minutes
  Insensitivity towards cold. Testing will start 10 minutes after end of LA infusion and continue every 5 minutes until onset is apparent.
Onset of motor nerve block | 10-180 minutes
  Paresis or paralysis of ankle dorsiflexion. Testing will start 10 minutes after end of LA infusion and continue every 5 minutes until onset of sensory nerve block is apparent.
Degree of sensory nerve block | 1-24 hours
  Grading system using a 4-level scale and compared to the contralateral leg: 1) normal; 2) different; 3) warmth; 4) no sensation. Testing will start after onset of sensory nerve block and will be done in intervals of 60 minutes hereafter and continue until return of normal sensation.
Degree of motor nerve block | 1-24 hours
  Grading system using a 3-level scale and compared to the contralateral leg: 1) normal; 2) paresis; 3) paralysis. Testing will start after onset of sensory nerve block and will be done in intervals of 60 minutes hereafter and continue until return of normal sensation.

CONTACTS AND LOCATIONS:
Overall Officials: Claus B Christiansen, MD, Principal Investigator — Nordsjaellands Hospital
Locations (1):
- Nordsjællands Hospital, Hillerød, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Christiansen CB, Madsen MH, Molleskov E, Rothe C, Lundstrom LH, Lange KHW. The effect of ropivacaine concentration on common peroneal nerve block duration using a fixed dose: A randomised, double-blind trial in healthy volunteers. Eur J Anaesthesiol. 2020 Apr;37(4):316-322. doi: 10.1097/EJA.0000000000001112. PMID 31789898